CLINICAL TRIAL: NCT03329300
Title: Using Executive Function to Predict Outcomes and Adherence in Family-based Behavioral Weight Management
Brief Title: Cognitive Aspects of Response to Treatment for Weight-related Health to Improve Eating and Exercise Earlier in Life
Acronym: CARTWHEEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Nutrition Obesity Research Center (Other)
Responsible Party: Principal Investigator, Marissa Gowey, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P30DK056336-16-PF-001; P30DK056336-16 (NIH)
Record Dates: First submitted 2017-10-25; First posted 2017-11-01 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-01

CONDITIONS: Pediatric Obesity; Executive Function
Keywords: Pediatric Obesity; Executive Function; Behavioral Intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): Family-based Behavioral Treatment (FBT)
  Interventions: Behavioral: Family-based Behavioral Treatment (FBT)

INTERVENTIONS:
Behavioral: Family-based Behavioral Treatment (FBT) — Family-based behavioral treatment (FBT) involves working with children and caregivers to modify diet and physical activity using behavioral strategies such as problem solving, goal setting, and self-monitoring. Children and caregivers will meet in group format on a weekly basis for 6 months. There will be 24 group session total, covering a variety of topics including nutrition, physical activity, and other aspects of health and wellness.

SUMMARY:
We plan to examine whether child and parental cognitive/executive function predict body composition outcomes and adherence to a 6-month protocol of Family-Based Behavioral Treatment (FBT), for pediatric obesity. Our objectives are to: (1) examine the effects of parent and child complex cognitive functions on treatment outcomes and adherence in a 6-month FBT program for obesity in a diverse group of children aged 8-12 (total of 16 child-parent pairs), and (2) examine the strength of the relationship between parent and child cognitive function. We hypothesize that children with poorer executive function, and those who have parents with poorer executive function, will have poorer body composition and adherence outcomes.

DETAILED DESCRIPTION:
Baseline assessments will include child and parent demographic data, medical history, and cognitive functioning, along with anthropometric measures such as height, weight, and body composition. Those who complete baseline assessments will be enrolled in one of two groups of family-based treatment on after-school evenings (8 pairs in each group; total of 16 child-caregiver pairs). A total of 24 weekly treatment sessions lasting up to 90 minutes each will be held over 6 months. Family-based behavioral treatment is a manualized, group intervention for children with obesity and their caregivers that incorporate participant-driven goal-based changes in diet and physical activity, and a variety of interactive educational session topics and behavioral support for reaching goals. A private weigh-in for children and caregivers will be conducted at each session. Sessions will begin with check-in with each family about weekly goal progress, after which the caregivers and children will split into separate groups for session-specific content including educational material tailored to nutrition, eating, and activity. The final portion of group session will involve children and caregivers merging in one group to share learning experiences and engage in collaborative goal-setting for the upcoming week(s). After the six month family-based behavioral intervention, baseline measures will be reassessed as well as overall program adherence. Program adherence will be evaluated using weekly program attendance and the number of days dietary/physical activity self-monitoring logs were completed.

ELIGIBILITY:
Inclusion Criteria:

1. Have a BMI ≥ 85th percentile
2. Are ≥8 and ≤12 years old at the beginning of treatment
3. Can read, write, and speak English, along with their parent
4. Plan to stay living within the local area during the study period
5. Have a consenting parent who can commit to all study procedures and provide reliable travel.

   * Siblings will be eligible for study inclusion if they meet the above criteria and will be allowed to use the same participating parent (sibling effects would then be addressed in statistical analyses).

Exclusion Criteria:

1. Have been diagnosed with a medical condition and/or are taking medication known to affect appetite/weight
2. Are currently participating in a formal weight management program beyond their usual medical care or have a parent participating in a formal weight management program
3. Have been diagnosed with an intellectual disability or traumatic brain injury
4. Have medical contraindications to physical activity.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Gowey, PhD, Principal Investigator — University of Alabama at Birmingham Department of Pediatrics
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Children; Parents/Caregivers: Family-based Behavioral Treatment (FBT)
  Family-based Behavioral Treatment (FBT): Family-based behavioral treatment (FBT) involves working with children and caregivers to modify diet and physical activity using behavioral strategies such as problem solving, goal setting, and self-monitoring. Children and caregivers will meet in group format on a weekly basis for 6 months. There will be 24 group session total, covering a variety of topics including nutrition, physical activity, and other aspects of health and wellness.
Period: Overall Study
Arm/Group | Children | Parents/Caregivers
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Children; Parents/Caregivers: There was one group of FBT participants comprised of parent/caregiver and child dyads. Separated for reporting of results only.
- Total: Total of all reporting groups
Arm/Group | Children | Parents/Caregivers | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (1.6) | 42.3 (8.9) | 26.21 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 5 | 6 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34
Child Body Fat Mass (DXA) [Mean (Standard Deviation); unit: %bf tblh (total body less head)] — Population: DXA scans were not performed on parents/caregivers
  %bf tblh (total body less head)
    number analyzed (Participants) | 17 | 0 | 17
    (all) | 48.8 (5.34) |  | 48.8 (5.34)
Child Body Mass Index [Mean (Standard Deviation); unit: Z-score] — Body mass index z-scores are measures of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Negative numbers indicate BMI values lower than the mean and positive numbers indicate BMI values higher than the mean. Population: Only child BMI is reported as a zscore
  Z-score
    number analyzed (Participants) | 17 | 0 | 17
    (all) | 2.41 (0.36) |  | 2.41 (0.36)
Parent Body Mass Index [Mean (Standard Deviation); unit: BMI Percentile] — Population: Only parent/caregiver BMI is reported as percentile
  BMI Percentile
    number analyzed (Participants) | 0 | 17 | 17
    (all) |  | 37.2 (12.6) | 37.2 (12.6)
Height [Mean (Standard Deviation); unit: cm] | 149.24 (7.27) | 163.35 (4.91) | 156.30 (9.41)
Weight [Mean (Standard Deviation); unit: kg] | 74.67 (20.11) | 98.20 (32.44) | 86.44 (29.14)
Executive Functioning [Mean (Standard Deviation); unit: t-score] — BRIEF Global Executive Composite, T-score:
  T-scores have a population mean of 50 and a standard deviation of 10.
  Higher scores indicate greater executive dysfunction. Corresponding T-scores and percentiles based on age and sex are assigned using raw scores. A score of 65 or above on any scale or index suggests potential clinical impairment (Gioia et al., 2000).
  t-score | 52.12 (11.11) | 52.71 (10.7) | 52.41 (10.74)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Child Body Fat Mass at 6 Months
Description: Dual-energy X-ray Absorptiometry (DXA)
Time Frame: Baseline to 6 months
Population: DXA scans were not performed on parents.caregivers.
Measure: Mean (Standard Deviation); unit: %bf tblh (total body less head)
Arm/Group | Children | Parents/Caregivers
Number analyzed (Participants) | 12 | 0
%bf tblh (total body less head) | -.96 (3.71) |

2. Secondary Outcome: Adherence to Treatment (Number of Contact Hours)
Description: The number of contact hours participant was exposed to treatment
Time Frame: Baseline to 6 months
Population: Assessed on the dyad level
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All Participants
Number analyzed (Participants) | 17
hours | 11.48 (10.49)

3. Secondary Outcome: Adherence to Treatment (Completed Days of Self-monitoring)
Description: The number of completed days of diet/activity self-monitoring using the USDA SuperTracker software, defined by ≥2 meals and exercise minutes recorded daily.
Time Frame: Baseline to 6 months
Population: Data were not collected; USDA Supertracker software was discontinued and thus not able to be used to collect data as planned.
Arm/Group | Children | Parents/Caregivers
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Child Height
Description: Height will be measured to the nearest 0.1 cm with a Seca 213 portable stadiometer.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Child Weight
Description: Weight will be measured to the nearest 0.1 kg with a Tanita SC-240 bio-electrical impedance (BIA) analyzer and standard scale.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Child Body Mass Index
Description: Body mass index z-scores are measures of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean.
  Change in child BMI z-score was calculated by subtracting child BMI z-score at 6 months from child BMI z-score at baseline. Negative scores indicate that BMI z-score decreased across the 6 month treatment period (i.e., better outcome), whereas positive scores indicate that BMI z-score increased from 0 to 6 months (i.e., worse outcome).
Time Frame: Baseline to 6 months
Population: Parent/caregiver BMI not reported as zscore
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Children | Parents/Caregivers
Number analyzed (Participants) | 13 | 0
z-score | -.05 (.05) |

7. Other Pre Specified Outcome: Parent/Guardian Height
Description: Height will be measured to the nearest 0.1 cm with a Seca 213 portable stadiometer.
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Parent/Guardian Weight
Description: as for outcome 5
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Parent/Guardian Body Mass Index
Description: Parent/guardian height and weight will be used together to determine BMI (kg/m^2). Raw BMI score at 6 months was subtracted from raw BMI score at baseline to calculate the change in BMI score from 0 to 6 months (i.e., treatment duration). Negative scores indicate a decrease in BMI (i.e., better outcome) whereas positive scores indicated an increase in BMI (i.e., worse outcome) from baseline to 6 months.
Time Frame: Baseline to 6 months
Population: Child BMI change not calculated using raw scores.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Children | Parents/Caregivers
Number analyzed (Participants) | 0 | 13
kg/m^2 |  | -.48 (1.02)

10. Other Pre Specified Outcome: Change in Executive Functioning - Inhibitory Control
Description: Performance-based EF was tested using the NIH Toolbox Cognitive Battery. NIH Toolbox T-scores were used (Mean=50, Standard deviation=10). Change in EF was calculated by subtracting the T-score at 6 months from the T-score at baseline. Positive change scores indicate an improvement in EF from baseline to 6 months, whereas negative change scores indicate a decline in EF from baseline to 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children | Parents/Caregivers
Number analyzed (Participants) | 10 | 10
t-score | 3.3 (5.43) | -2.00 (5.39)

11. Other Pre Specified Outcome: Change in Executive Functioning - Working Memory
Description: as for outcome 10
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children | Parents/Caregivers
Number analyzed (Participants) | 10 | 10
t-score | .40 (6.36) | 4.30 (6.75)

12. Other Pre Specified Outcome: Change in Executive Functioning - Cognitive Flexibility
Description: as for outcome 10
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Children | Parents/Caregivers
Number analyzed (Participants) | 10 | 10
t-score | 5.40 (7.26) | 6.40 (12.81)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Children | Parents/Caregivers
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03329300/Prot_SAP_000.pdf